CLINICAL TRIAL: NCT05855447
Title: Intercostal and Quadriceps Femoris Muscles Oxygenation During Exercise in Patient With Fibrosing Interstitial Lung Diseases
Brief Title: Muscles Oxygenation During Exercise in Fibrosing Interstitial Lung Diseases
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Fibrozan_Moxy_1
Record Dates: First submitted 2023-04-17; First posted 2023-05-11 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-02

CONDITIONS: Lung Diseases, Interstitial; Exercise, Compulsive; Oxygen Deficiency
Keywords: Oxygen Consumption; Interstitial Lung Diseases; Exercise
MeSH Terms: conditions — Lung Diseases, Interstitial; Compulsive Exercise; Hypoxia; Motor Activity | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fibrosing Lung Disease Group: It will consist of 36 patients diagnosed with ILD. The patients whose demographic information such as age, height and weight will be questioned will then be evaluated with a desktop spirometer, peripheral muscle strength measurement with a digital myometer, and functional capacity with a 6MWT. The Moxy device, which is a NIRS, will be attached to the upper leg (the vastus lateralis of the quadriceps muscle) and the rib (intercostal muscles) with a silk patch, and the oxygenation of the muscles here will be measured during the 6MWT. In addition, fatigue status will be evaluated with the Modified Borg Scale.
  Interventions: Other: NIRS device usage during 6MWT; Other: Peripheral Muscle Strength Measurement; Other: Pulmonary Function Test

INTERVENTIONS:
Other: NIRS device usage during 6MWT — It will be performed by placing a traffic cone as the sign of the turning point in a straight 30 meter long corridor, after patients have rested for a sufficient time (> 30 minutes) by sitting in a chair. Participants will be asked to walk as fast as possible but without running along the corridor within 6 minutes. Before and after the test, the patient's fatigue and dyspnea conditions will be questioned using the Modified Borg Scale and blood pressure using a digital sphygmomanometer, and saturation and pulse measurement will be evaluated using finger pulse oximetry before, during and after the test. During the 6-minute walk test, the muscle oxygenation of the patients and the amount of muscle oxygen will be measured using Moxy (Fortiori Design LLC, Minnesota, USA) brand NIRS technology. During the walking test, the change in intramuscular oxygenation will be monitored and recorded with the company's software program.
Other: Peripheral Muscle Strength Measurement — The muscle strength of shoulder flexors, abductors, elbow flexors, hip flexors, abductors, and knee extensors will be evaluated using a Lafayette® 01165 model electronic hand dynamometer. The force measurement will be repeated 3 times and it will be requested to maintain muscle strength against the dynamometer for at least 5 seconds in each trial. The best value out of 3 test results will be recorded
Other: Pulmonary Function Test — Pulmonary Function Test (PFT) with desktop type spirometry for FVC (Forced Vital Capacity), Forced expiratory flow rate (FEV1), FEV1/FVC.

SUMMARY:
The type of this study is an observational prospective study. It will be done to determine the oxygenation status of the intercostal muscles and quadriceps femoris muscle during exercise in patients with fibrosing lung and to examine its relationship with exercise capacity, respiratory functions and respiratory muscle strength. The main questions that the study aims to answer are:

* Question 1: Do changes in muscle oxygenation during exercise affect respiratory functions in patients with Fibrosing Lung?
* Question 2: Do changes in muscle oxygenation during exercise affect exercise capacity in patients with Fibrosing Lung?

Participants; demographic information such as age, height, weight will be questioned. Respiratory functions will be evaluated with a desktop spirometer, peripheral muscle strength measurement will be evaluated with a digital myometer, and functional capacity will be evaluated with a 6-minute walk test (6MWT). The Moxy device, which is a non-invasive near-infrared spectroscopy (NIRS), will be attached to the upper leg (the vastus lateralis of the quadriceps muscle) and the rib (intercostal muscles) with a silk patch, and the oxygenation of the muscles here will be measured during the 6-minute walking test. In addition, fatigue status will be evaluated with the Modified Borg Scale.

DETAILED DESCRIPTION:
Interstitial Lung Disease (ILD); It constitutes a heterogeneous group of approximately 200 diseases with acute or chronic course that affect the lung diffusely and cause varying degrees of inflammation, fibrosis and structural deterioration in the lung parenchyma. Clinical features of ILD include exercise-induced dyspnea, exercise-induced hypoxemia, progressive skeletal muscle weakness, and impaired exercise tolerance. The main symptoms of fibrosis are progressive decreases in forced vital capacity (FVC) and diffusing capacity of the lung for carbon monoxide (DLCO). Restriction of pulmonary ventilation leads to respiratory failure, which is exacerbated by capillary destruction and decreased alveolar blood flow resulting from hypoxic vasoconstriction.

Exercise intolerance is a key feature of ILD and is usually associated with significant dyspnea on exertion. Exercise limitation in ILD is related to altered respiratory mechanics, impaired gas exchange, and circulatory limitation. Evidence suggests that pulmonary rehabilitation can provide significant benefits in patients with ILD. Daily use of corticosteroids for >1 year significantly reduces muscle function in patients with chronic respiratory disease. Muscle size, strength, and functional outcomes were evaluated in ILD patients. Decreased quadriceps strength and endurance were seen in patients with fibrotic idiopathic interstitial pneumonia compared to healthy controls. Compared to the upper extremity, more atrophy and weakness were found in the lower extremity muscles. Therefore, exercise training is a critical component of pulmonary rehabilitation. The effect of exercise on blood oxygenation has been little studied in ILD patients, and the few data available in the literature are conflicting.

In the studies conducted, there are studies stating that there is a positive improvement in blood biochemistry as a result of an acute exercise, as well as a change with chronic exercises. An important goal of hemodynamic monitoring is the early detection of inadequate tissue perfusion and oxygenation. The use of simple, non-invasive monitoring techniques has the advantage of facilitating earlier initiation of therapy. Near-infrared spectroscopy (NIRS) is a noninvasive measurement instrument that does not impair skin integrity, allowing the measurement of muscle hemoglobin-oxygen saturation (StO2) during exercise. There are few studies in the literature where muscle oxygenation was measured with the NIRS device. According to the results of our literature review, our study will be the first study to examine muscle oxygenation in fibrosing lung patients.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-75.
* Have a diagnosis of fibrosing interstitial lung disease diagnosed according to the clinical diagnostic criteria of the American Thoracic and European Respiratory Societies (ATS-ERS).
* Presence of dyspnea on exertion Stable clinical state at the time of admission without infection or exacerbation in the previous 4 weeks.
* Ability to use a smart phone.

Exclusion Criteria:

* Patients with severe comorbid diseases, unstable coronary artery disease, collagen vascular diseases and needing high flow oxygen therapy (˃ 3-4 L \min).
* History of effort-related syncope or any comorbidity (such as severe orthopedic or neurological deficits or unstable heart disease) that precludes exercise training.
* Participating in a pulmonary rehabilitation program within the past 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample of the study will consist of male and female patients between the ages of 18-75 who have been diagnosed with Fibrosing Lung Disease (Interstitial Lung Disease) in Istanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Relative Muscle Oxygenation Changes with Moxy Muscle Oxygenation Monitor (SmO2) | Through study completion, an average of 1 year
  The measurement will be made in the dominant lower extremity, and the device will be measured by placing the device at a distance of 5 cm from the anterior superior reference point of the spina iliaca to the mid-thigh region of the midpoint of the patella, the intersection of the sixth and eighth intercostal spaces, and the anterior axillary line. Relative muscle oxygenation changes (SmO2) and total hemoglobin concentration according to the modified Beer-Lambert Law formula (SmO2 = (Hb +) by comparing the measured light intensities with a pre-computed data set obtained by a Monte Carlo (MC). O2Mb) ÷ [(O2Hb + O2Mb) + (HHb + HMb)]) percent SmO2 concentration is determined by the diffusion of light in tissue layers.
Total Hemoglobin Concentration with Muscle Oxygenation Monitor (SmO2) | Through study completion, an average of 1 year
  The measurement will be made in the dominant lower extremity, and the device will be measured by placing the device at a distance of 5 cm from the anterior superior reference point of the spina iliaca to the mid-thigh region of the midpoint of the patella, the intersection of the sixth and eighth intercostal spaces, and the anterior axillary line. Relative muscle oxygenation changes (SmO2) and total hemoglobin concentration according to the modified Beer-Lambert Law formula (SmO2 = (Hb +) by comparing the measured light intensities with a pre-computed data set obtained by a Monte Carlo (MC). O2Mb) ÷ [(O2Hb + O2Mb) + (HHb + HMb)]) percent SmO2 concentration is determined by the diffusion of light in tissue layers.

SECONDARY OUTCOMES:
Digital Muscle Strength Measurement for Peripheral Muscle Strength | Before 6MWT
  Muscle strength of shoulder flexors, abductors, elbow flexors, hip flexors, abductors, and knee extensors will be evaluated. The test will be done by Lafayette brand digital muscle strength meter.
Pulmonary Function Test for FVC | Before 6MWT
  Pulmonary function test will be performed with desktop type spirometry. The FVC value will be calculated.
Pulmonary Function Test for FEV1 | Before 6MWT
  Pulmonary function test will be performed with desktop type spirometry. The FEV1 value will be calculated.
Pulmonary Function Test for FEV1/FVC | Before 6MWT
  Pulmonary function test will be performed with desktop type spirometry. The FEV1/FVC value will be calculated.
Maximal Inspiratory Muscle Strength | Before 6MWT
  Pulmonary function test will be performed with desktop type spirometry. The Maximal Inspiratory Pressure value will be calculated.
Maximal Expiratory Muscle Strength | Before 6MWT
  Pulmonary function test will be performed with desktop type spirometry. The Maximal Expiratory Pressure value will be calculated.
Fatigue measured with the Modified Borg Scale | Before 6MWT
  Fatigue severity will be measured with the Modified Borg Scale. In the scale, the severity of fatigue is measured with a score between 0 and 10 points. On this scale, 0 point defines the best condition in terms of fatigue, and 10 points the worst.
Dyspnea measured with the Modified Borg Scale | Before 6MWT
  Dyspnea severity will be measured with the Modified Borg Scale. In the scale, the severity of dyspnea is measured with a score between 0 and 10 points. On this scale, 0 point defines the best condition in terms of dyspnea, and 10 points the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Esra PEHLİVAN, Assoc. Prof., Principal Investigator — Saglik Bilimleri Universitesi; Erdoğan ÇETİNKAYA, Prof. Dr., Study Director — Saglik Bilimleri Universitesi; Zeynep Betül ÖZCAN, M. Sc., Study Chair — Saglik Bilimleri Universitesi; Fulya Senem KARAAHMETOĞLU, M. Sc., Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- SBU Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)